CLINICAL TRIAL: NCT06211218
Title: Application of Deep Learning for Screening Multiple Corneal Diseases
Brief Title: Artificial Intelligence for Screening of Multiple Corneal Diseases
Status: Recruiting | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2023083
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Deep Learning; Corneal Disease; Screening
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cornea diseases diagnosed by artificial intelligence algorithm
  Interventions: Diagnostic Test: Cornea diseases diagnosed by artificial intelligence algorithm

INTERVENTIONS:
Diagnostic Test: Cornea diseases diagnosed by artificial intelligence algorithm — An artificial intelligence algorithm was applied to diagnose cornea diseases from slit-lamp images.

SUMMARY:
This study developed a deep learning algorithm based on anterior segment images and prospectively validated its ability to identify corneal diseases.The effectiveness and accuracy of this algorithm was evaluated by sensitivity, specificity, positive predictive value, negative predictive value, and area under curve.

ELIGIBILITY:
Inclusion Criteria:

1. The quality of slit-lamp images should clinical acceptable.
2. More than 90% of the slit-lamp image area including three main regions (sclera, pupil, and lens) are easy to read and discriminate.

Exclusion Criteria:

1）Insufficient information for diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is derived from an anonymous database that contains health examination results of the general population.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-12-06 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
Area under curve | 1 week
  We used the receiver operating characteristic (ROC) curve and area under curve to examine the ability of this artificial intelligence algorism recognition and classification of corneal diseases.
Sensitivity and specificity | 1 week
  We used sensitivity and specificity to examine the ability of this artificial intelligence algorism recognition and classification of corneal diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Prof, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided